CLINICAL TRIAL: NCT06021652
Title: Feasibility, Adoption and Efficacy of A Virtual Reality Smoking Cessation Program for Patients Undergoing Lung Cancer Screening: A Pilot Trial
Brief Title: Feasibility, Adoption and Efficacy of A Virtual Reality Smoking Cessation Program for Patients Undergoing Lung Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: MindCotine (Unknown)
Responsible Party: Principal Investigator, Sara Ghandehari, Professor of Medicine, Division of Pulmonary and Critical Care Medicine, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002746
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco use; Virtual Reality; Smoking cessation
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants electing to participate in the virtual reality based smoking cessation platform
  Interventions: Device: MindCotine Virtual reality
- Control (No Intervention): Those utilizing standard of care smoking cessation therapies

INTERVENTIONS:
Device: MindCotine Virtual reality — Virtual reality platform
  Arms: Virtual Reality

SUMMARY:
Lung cancer is the second most common cancer and the leading cause of cancer related deaths in the United States (US . Tobacco use is the leading cause of lung cancer and tobacco control continues to be the primary method of lung cancer prevention. Smoking cessation interventions (SCIs) are strongly recommended by screening guidelines and have a class A recommendation by the United States Preventive Services Task Force. Currently, a variety of smoking cessation interventions exist, and evidence suggests that pharmacotherapy, such as nicotine replacement therapy, in combination with behavioral interventions is more effective than either intervention alone. Many individuals, however, prefer not to use or are unable to use pharmacotherapy. A variety of behavioral interventions exist to aid in smoking cession. Recently, virtual reality (VR) has emerged as a possible tool to conduct behavior interventions. Previous research has demonstrated that use of VR can improve patient engagement in a variety of chronic disease interventions. Little is known however about the feasibility and adoption of VR in smoking cessation, especially among individuals at high risk for lung cancers. VR based platforms utilize 'cue exposure therapy'. Given that cravings are often triggered by external factors, or cues, cue exposure therapy exposes individuals to repeated drug-related cues and provides them with tools to eliminate cue-induced cravings. Given the inability for all individuals to use pharmacotherapy there remains a critical need to improve adherence to and efficacy of behavioral interventions for smoking cessation. To address this unmet need, the investigators propose, as pilot study, to enroll patients undergoing routine lung cancer screening and who are not interested in or cannot take pharmacologic therapies for smoking cession, to participate in VR based smoking cessation therapy.

DETAILED DESCRIPTION:
The purpose of this study is to assess the adoption rate of VR smoking cessation intervention (MindCotine app) in those who are at risk for lung cancer and are participating in a lung cancer screening program.

The investigators will enroll 20 individuals. 10 of whom elect to participate in the VR program and 10 of whom are using standard of care smoking cessation methods.

The study duration is 90 days after completion of the MindCotine VR program. The MindCotine program consists of a 8-week training stage, and includes audiovisual content, cognitive behavioral therapy based self-reflective questions, setting a quit date, and notifications. The audio-visual content includes formal mindfulness exercises involving breathing techniques, body awareness, thought recognition, emotions, and smoking impulses. VR therapy exercises include the following topics: The Act of Smoking; RAIN meditation; Stress at work; Bodily sensations; Deep emotions; Nicotine anonymous; Alcohol as a trigger. Each content consists of a 2 minute animated environment to induce meditative states of mind, 6 minutes of exposure with real people, and 2 more minutes of an animated environment to induce a meditative mindset.

Participants will be surveyed at baseline, 1 day after the completion of the 8 week VR program and again 90 days after the completion of the VR program.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand informed consent
* Easy access to personal smartphone o Male or female adults who are at high risk for lung cancer and are enrolled in the Cedars-Sinai lung cancer screening program A: Based on USPSTF guidelines: Age 50-80 with 20 or greater pack-year smoking story who continue to smoke B: Based on National Comprehensive Cancer Network (NCCN) guidelines but do not meet the USPSTF guidelines, age 50-unlimited

Exclusion Criteria:

* Persons with photosensitive epilepsy will be excluded; flashing scenes in the virtual reality can trigger seizures.
* Any records flagged "break the glass" or "research opt-out."
* Persons who are unable to use smart phone or have a smartphone that is not compatible with a virtual reality app. The app is currently available in English and Spanish, and those who are not fluent in speaking and reading English or Spanish are excluded from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 1 year
  Ability to recruit our target number of participants during the study period
Adoptability | 1 year
  Adoption rate will be assess as those who complete at least 75% of the VR content compared to the total persons enrolled in the study

SECONDARY OUTCOMES:
efficacy of smoking cessation | 1year
  percentage of persons who stopped smoking during the course of the study in the VR group compared to controls

IPD SHARING:
Plan to Share IPD: No